CLINICAL TRIAL: NCT00046787
Title: Phase II Study to Determine the Efficacy of OSI-211 (Liposomal Lurtotecan) Given on Days 1, 2 & 3 Every 3 Weeks in Patients With Recurrent Small Cell Lung Cancer
Brief Title: Efficacy and Safety Study of OSI-211 (Liposomal Lurtotecan) to Treat Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110-12
Record Dates: First submitted 2002-10-03; First posted 2002-10-04 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: SCLC; Carcinoma, Small Cell
Keywords: Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Small Cell; Small Cell Lung Carcinoma | interventions — lurtotecan

INTERVENTIONS:
Drug: OSI-211 (Liposomal Lurtotecan)

SUMMARY:
The purpose of this study is to determine whether OSI-211 (Liposomal Lurtotecan) is an effective and safe treatment for patients with recurrent small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed recurrent small cell lung cancer.
* One prior treatment of chemotherapy.
* At least three weeks since last chemotherapy treatment and recovery from any related side effects.
* At least three weeks since last chest radiotherapy and at least 10 days since head irradiation and recovery from acute side effects.
* At least one target tumor less than or equal to 20 mm (or less than or equal to 10 mm on spiral CT-scan).
* If a patient has had previous documented Central Nervous System (CNS) involvement, only controlled disease is acceptable.

Exclusion Criteria:

* Superior vena cava syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47
Dates: Start 2002-09; Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Baptist Hospital Regional Cancer Ctr., Knoxville, Tennessee
  - Vanderbilt Clinical Trials Office, Nashville, Tennessee
- United Kingdom (6):
  - Nottingham City Hospital, Nottingham, Nottinghamshire
  - Clatterbridge Centre for Oncology, Bebington, Wirral
  - Aberdeen Royal Infirmary, Aberdeen
  - Guys Hospital, London
  - Christie Hospital, Manchester
  - Northern Centre for Cancer Research, Newcastle General Hospital, Newcastle upon Tyne